CLINICAL TRIAL: NCT02608385
Title: Phase I Study of PD1 Blockade by Pembrolizumab With Stereotactic Body Radiotherapy in Advanced Solid Tumors
Brief Title: Study of PD1 Blockade by Pembrolizumab With Stereotactic Body Radiotherapy in Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB15-1130
Record Dates: First submitted 2015-11-09; First posted 2015-11-18 (Estimated); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Solid Tumor
MeSH Terms: interventions — Radiosurgery; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dose Escalation Cohort (Experimental): Patients will be enrolled to receive specific doses of radiation (stereotactic body radiotherapy) given over 1 week followed by treatment with pembrolizumab. Pembrolizumab dosing will continue for up to 2 years or until patients have disease progression or unacceptable side effects. Enrollment will continue until best safe dose of SBRT is determined for each organ type.
  Interventions: Radiation: Stereotactic body radiotherapy (SBRT); Drug: Pembrolizumab
- Large Volume Tumors Cohort (Experimental): Patients with large tumors will be enrolled and their tumors will be partially treated with (stereotactic body radiotherapy) given over 1 week followed by treatment with pembrolizumab. Pembrolizumab dosing will continue for up to 2 years or until patients have disease progression or unacceptable side effects.
  Interventions: Radiation: Stereotactic body radiotherapy (SBRT); Drug: Pembrolizumab
- Oligometastatic Cohort (Experimental): Patients with few tumors (4 or less) will be enrolled and their tumors treated with (stereotactic body radiotherapy) given over 1 week followed by treatment with pembrolizumab. Pembrolizumab dosing will continue for up to 2 years or until patients have disease progression or unacceptable side effects.
  Interventions: Radiation: Stereotactic body radiotherapy (SBRT); Drug: Pembrolizumab

INTERVENTIONS:
Radiation: Stereotactic body radiotherapy (SBRT) — Patients will receive 3 or 5 doses of SBRT to the chosen metastases.
Drug: Pembrolizumab — Pembrolizumab (200 mg) given every 3 weeks.
  Other Names: Keytruda

SUMMARY:
Phase I to determine safety of combining stereotactic body radiotherapy (SBRT) with pembrolizumab in patients with advanced solid tumors. The study will determine safe doses of radiation by organ site when used together with pembrolizumab. The study will also provide the opportunity to evaluate changes in the tumor caused by SBRT.

The study will include 2 expansion cohorts:

* Partially Irradiated Large Volume Tumors Cohort: Patients with at least one lesion greater than 65cc amenable to SBRT followed by pembrolizumab.
* Oligometastatic Cohort: Patients with limited metastatic disease (4 or fewer lesions)

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent/assent for the trial.
* Aged 18 years or older
* Have a histologically confirmed advanced solid tumor for which curative treatment is not available.
* Have undergone all appropriate standard of care treatment options (in the opinion of the treating investigator). Patients with NSCLC must have undergone EGFR and ALK testing and have received appropriate initial therapy.
* Have measurable disease based on RECIST 1.1 including at least two tumor lesions that meet criteria for multi-organ site ablative radiation therapy (MOSART) SBRT radiation.

  * 0.25 cc to 65 cc of viable tumor (i.e. primary disease or metastases) approximately 5cm in maximal dimension. Tumors larger than 65 cc can be partially treated. Patients accruing to the expansion cohort for partially irradiated large tumors must have at least one site of disease >65cc.
  * Metastases located in lung, liver, mediastinal/cervical node, Spinal/Paraspinal, Osseous, abdominal-pelvic (lymph node/adrenal gland)
* For biopsy patients: Be willing to undergo repeat biopsy of a tumor lesion before treatment and after radiation. Subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may be exempted from this requirement after consultation with the Principal Investigator.
* Have a performance status of 0 or 1 on the ECOG Performance Scale.
* Demonstrate adequate organ function

  * Absolute neutrophil count (ANC) ≥ 1,500 /mcL
  * Platelets ≥ 100,000 / mcL
  * Hemoglobin ≥ 8 g/dL
  * Serum creatinine OR Measured or calculateda creatinine clearance ≤ 1.5 X upper limit of normal (ULN) OR ≥ 50 mL/min for subject with creatinine levels > 1.5 X institutional ULN
  * Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN
  * AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases
  * Albumin ≥ 3.0 mg/dL
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.
* Have an investigator determined life expectancy of at least 6 months.

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy at a dose of >10 mg Prednisone daily or equivalent at time of first dose of trial treatment.
* Has a known history of active TB (Bacillus Tuberculosis)
* Hypersensitivity to pembrolizumab or any of its excipients.
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from side effects due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

  * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
  * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has known history of non-infectious pneumonitis that required steroids or active pneumonitis.
* Has evidence of interstitial lung disease.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment.
* If known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA qualitative is detected) then patient is not eligible for cohorts including SBRT to liver lesions.
* Has received a live vaccine within 30 days of planned start of study therapy.

  * Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed, however intranasal influenza vaccines are live attenuated vaccines and are not allowed.
* Has had prior radiation therapy (defined as >10% of prior prescription dose) to the area planning to be treated with SBRT

Additional Criteria for Expansion Cohorts:

* Partially Irradiated Large Volume Tumors Cohort

  * In addition to the criteria above, patients must have at least one lesion >65cc (~5cm diameter sphere) that is amenable to partial tumor irradiation.
* Oligometastatic disease

  * In addition to the criteria above, patients must have disease limited to 4 total lesions or less, all of which are amenable to SBRT. Patients with oligometastatic disease at presentation or oligorecurrent disease are eligible. Patients who had more than 4 sites of disease previously, but had a complete response at other sites and limited progressive disease to 4 sites are eligible for participation. Partial tumor irradiation for lesions >65cc is permitted in this expansion cohort.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2015-12; Primary Completion 2022-04-01 (Actual); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Recommended stereotactic body radiotherapy (SBRT) dose in combination with pembrolizumab. | 3 Months
  To determine the recommended SBRT dose to various metastatic locations in patients with advanced solid tumors, and specifically in the lung in patients with NSCLC, in conjunction with pembrolizumab treatment.
  Each metastasis targeted with SBRT will be assigned to one of the seven "Metastasis Locations". Patients will receive 3 or 5 fractions of radiation as determined by the location of the metastases to be irradiated.
  Exact logistic regression 13 analyses will be conducted to model the probability of DLT as a function of site dose, number of metastatic sites, and cumulative body radiation. These analyses will be conducted separately for each site using all patients with lesions at that site. If these analyses suggest a high (>=33%) probability of toxicity for a particular combination of predictors, dose recommendations may be modified

SECONDARY OUTCOMES:
Rate of side effects | 3 Months
  To estimate rates of ≥ grade 3-4 adverse events, scored according to NCI CTCAE v. 4.0, by organ system
Rate of long term side effects | 24 Months
  Rates of long-term adverse events, scored according to NCI CTCAE v. 4.0,
Response rate | 24 Months
  Response rates will be tabulated with 90% confidence limits based on the binomial distribution.
Progression-free survival | 12 months
  Progression-free survival will be estimated using the Kaplan-Meier method.
Overall survival | 24 months
Local control of SBRT lesion | 12 months
Changes in tumor microenvironment caused by radiation treatment | 1 week
Effect of radiation and pembrolizumab on tumor control for lesions larger than 65cc | 12 months
Effect of combining radiation and pembrolizumab on local and distant tumor control | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Steven Chmura, M.D., Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Korpics MC, Onderdonk BE, Dadey RE, Hara JH, Karapetyan L, Zha Y, Karrison TG, Olson AC, Fleming GF, Weichselbaum RR, Bao R, Chmura SJ, Luke JJ. Partial tumor irradiation plus pembrolizumab in treating large advanced solid tumor metastases. J Clin Invest. 2023 May 15;133(10):e162260. doi: 10.1172/JCI162260. PMID 37183819